CLINICAL TRIAL: NCT07159074
Title: Repurposing Tc 99m Tilmanocept Imaging for Cardiac Sarcoidosis
Brief Title: Repurposing Tilmanocept for Cardiac Sarcoidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Foundation for Sarcoidosis Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO00117849
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Cardiac Sarcoidosis
MeSH Terms: interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tc 99m Tilmanocept SPECT CT imaging (Experimental): Participants with known cardiac sarcoidosis and a cardiac positron emission tomography (PET) imaging study showing active inflammation in the past 14 days or participants with a cardiomyopathy for which sarcoidosis has been excluded will undergo Single Photon Emission Computed Tomography (SPECT-CT) imaging after administration of Tc 99m Tilmanocept intravenously.
  Interventions: Drug: Tc 99m tilmanocept

INTERVENTIONS:
Drug: Tc 99m tilmanocept — 150 mcg containing 10 mCi of Tc 99m tilmanocept will be administered through an IV route of injection. SPECT-CT imaging will then be performed.

SUMMARY:
The purpose of this study is to see if Tc 99m Tilmanocept SPECT/CT imaging can be used to identify cardiac sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

Cohort 1:

1. The participant has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) or equivalent authorization before the initiation of any study-related procedures.
2. Women of reproductive potential must have a negative urine pregnancy test at the time of the study.
3. The participant is at least 18 years of age.
4. The participant has a histological diagnosis sarcoidosis and meets 2014 HRS, 2014 WASOG, or 2016 JCS criteria for cardiac sarcoidosis.
5. The participant has had a clinically indicated cardiac PET-CT showing cardiac activity in the past 14 days.
6. The participant has had a prior cardiac MRI with delayed enhancement in pattern consistent with cardiac sarcoidosis as defined in the AHA Scientific Statement on the Diagnosis and Management of Cardiac Sarcoidosis (2024).

Cohort 2:

1. The participant has provided written informed consent with HIPAA (Health Information Portability and Accountability Act) or equivalent authorization before the initiation of any study-related procedures.
2. Women of reproductive potential must have a negative urine pregnancy test at the time of the study.
3. The participant is at least 18 years of age.
4. Cardiac sarcoidosis has been clinically excluded.
5. The participant has an arrhythmogenic, non-ischemic cardiomyopathy defined as the presence of a cardiomyopathy with a history of recurrent (more than 1 episode) ventricular tachycardia, atrial arrhythmias, high grade AV block not due to ischemic heart disease

Exclusion Criteria:

1. The participant is pregnant or lactating.
2. The participant size or weight is not compatible with imaging per the investigator.
3. The participant has renal insufficiency as demonstrated by a glomerular filtration rate of < 30 mL/min.
4. The participant has hepatic insufficiency as demonstrated by ALT (alanine aminotransferase [SGPT]) or AST (aspartate aminotransferase [SGOT]) greater than 3 times the upper limit of normal.
5. The participant has any severe, acute, or chronic medical conditions and/or psychiatric conditions and/or laboratory abnormalities that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration that would deem the subject inappropriate for study participation.
6. The participant has a known allergy to or has had an adverse reaction to dextran exposure.
7. The participant has received an investigational product within 30 days prior to the Tc 99m tilmanocept administration (Day 0).
8. The participant has received any radiopharmaceutical within 7 days or 10 half-lives prior to the administration of Tc 99m tilmanocept (Day 0).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between the cardiac segments with tilmanocept uptake and the cardiac segments with fluorodeoxyglucose (FDG) uptake on cardiac PET-CT. For each imaging modality, a standard 17-segment cardiac model will be used. | At the time of the scan (Baseline)

SECONDARY OUTCOMES:
Correlation between TUVmax from tilmanocept imaging and SUVmax from FDG-PET imaging. | At the time of the scan (Baseline)
Correlation between the cardiac segments with tilmanocept uptake and the cardiac segments with hyperenhancement on cardiac MRI. For each imaging modality, a standard 17-segment cardiac model will be used. | At the time of the scan (Baseline)
Correlation of extracardiac sites with tilmanocept uptake and FDG uptake attributed to sarcoidosis. | At the time of the scan (Baseline)
Difference in percentage of segments with tilmanocept uptake in cohort 1 compared to cohort 2 | At the time of the scan (Baseline)
Adverse events, identified through clinical laboratory results (hematology, serum chemistry, vital signs). | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Karra, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No